CLINICAL TRIAL: NCT03103048
Title: Application of Different Techniques of Elastic Bandage: Quantification Electromyographic at the Isometric Effort of Flexor Muscle of Fist
Brief Title: Application of Different Techniques of Elastic Bandage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Principal Investigator, University of Mogi das Cruzes
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CAAE 64513617.3.0000.5497
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2017-04

CONDITIONS: Forearm Muscle Strain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): The tests will be performed in thirty days, session with lasting 15 minutes each, when all volunteers will be submitted in four measure tests: 1- Without bandages (start); 2 - With placebo; 3 - With bandage; 4 - With tensioned bandage.
  Interventions: Diagnostic Test: Without bandages; Diagnostic Test: With placebo; Diagnostic Test: With bandage; Diagnostic Test: With tensioned bandage
- Group 2 (Placebo Comparator): The tests will be performed in thirty days, session with lasting 15 minutes each, when all volunteers will be submitted in four measure tests: 1- Without bandages; 2 - With placebo (start); 3 - With bandage; 4 - With tensioned bandage.
  Interventions: Diagnostic Test: Without bandages; Diagnostic Test: With placebo; Diagnostic Test: With bandage; Diagnostic Test: With tensioned bandage
- Group 3 (Active Comparator): The tests will be performed in thirty days, session with lasting 15 minutes each, when all volunteers will be submitted in four measure tests: 1- Without bandages; 2 - With placebo; 3 - With bandage (start); 4 - With tensioned bandage.
  Interventions: Diagnostic Test: Without bandages; Diagnostic Test: With placebo; Diagnostic Test: With bandage; Diagnostic Test: With tensioned bandage
- Group 4 (Active Comparator): The tests will be performed in thirty days, session with lasting 15 minutes each, when all volunteers will be submitted in four measure tests: 1- Without bandages; 2 - With placebo; 3 - With bandage; 4 - With tensioned bandage (start).
  Interventions: Diagnostic Test: Without bandages; Diagnostic Test: With placebo; Diagnostic Test: With bandage; Diagnostic Test: With tensioned bandage

INTERVENTIONS:
Diagnostic Test: Without bandages — All volunteers will be held the grasping force measurements without application of elastic adhesive bandage or micropore
Diagnostic Test: With placebo — All volunteers will be held the grasping force measurements with application of micropore (placebo) on his forearm in both upper members
Diagnostic Test: With bandage — All volunteers will be held the grasping force measurements with application of bandage without tension in the forearm in both upper members
Diagnostic Test: With tensioned bandage — All volunteers will be held the grasping force measurements with application of bandage with twenty five percent tensioned on the forearm in both upper members

SUMMARY:
This study will be featured as a randomized controlled. As the dependent variable, was considered isometric grip manual force. As independent variable, the presence or absence of forearm bandage in the fist flexor region of the volunteers.

DETAILED DESCRIPTION:
This study is directed to the population of students at the University of Mogi das Cruzes (UMC), and will take part of this study forty volunteers, twenty men and twenty women, aged from eighteen and thirty-eight years old. Will be selected and included volunteers who do not do physical professional activity with upper members, which have no symptom of pain skeletal muscle in the upper members, which have not undergone any type of surgery in the region of the forearm and hand of both members. Will be excluded the volunteers who have injuries, joint injuries, neuromuscular disorder or those who have knowledge of own vestibular or neurological changes. Will also be excluded from study volunteers who do not agree to participate after reading and understanding of informed consent in accordance with resolution 466/12 of the National Ethics Committee and Research. The data acquisition interface will be acquired by an electromyography e a standard of strentgh will maintened in forty Newtons assured by an electronic dynamometer for tests of palmar prehension without and with bandages. The volunteers will not know what kind of intervention will pass. After each application before testing, their both forearms will be covered with a protection. The researcher and the volunteers will not know the tests order.

ELIGIBILITY:
Inclusion Criteria:

* Who do not do physical professional activity with upper members;
* Who have no symptom of pain skeletal muscle in the upper members;
* Who have not undergone any type of surgery in the region of the forearm and hand of both members;
* Consent form signed by the volunteer.

Exclusion Criteria:

* Having less than 18 years old;
* Having more than 38 years old;
* To present some compromise skeletal muscle in the upper members;
* Who do not want take part in the research;
* Who do not signed consent form as volunteer.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Efforts | 15 minutes
  Thru palmar prehension there will be data acquisition interface by an electromyography e a standard of strentgh maintened in 40 Newtons assured by an electronic dynamometer for tests of palmar prehension, with and without elastic adhesive bandages in the region of flexor muscle of fist.

CONTACTS AND LOCATIONS:
Overall Officials: Terigi A Scardovelli, Ph.D., Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Terigi Augusto Scardovelli, Mogi das Cruzes, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided